CLINICAL TRIAL: NCT07385560
Title: "The Importance of Adding Fenestration to Ultrasound-Guided Baker's Cyst Aspiration"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tutku naz bulut, Resident Physician, Department of Physical Medicine and Rehabilitation, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-24687290-604.01-1407310; E-24687290-604.01-1407310 (Other: Istanbul University-Cerrahpasa Ethics Committee)
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Baker Cyst; Fenestration; Musculoskeletal Ultrasound; Steroid Injection; OMERACT; Knee Osteoarthritis
Keywords: Baker's cyst; Knee osteoarthritis; Ultrasound-guided aspiration; Steroid injection; Lidocaine; Fenestration; OMERACT; WOMAC; Musculoskeletal ultrasound; Cyst recurrence; KOOS
MeSH Terms: conditions — Popliteal Cyst; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: "Two-arm, parallel-group, randomized controlled interventional study evaluating the clinical effects of adding fenestration to ultrasound-guided aspiration."
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants and investigators who perform evaluations are blinded to group assignment. The clinician performing the ultrasound-guided procedure is not involved in outcome assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspiration + Steroid-Lidocaine (Active Comparator): Ultrasound-guided aspiration of Baker's cyst followed by injection of corticosteroid and lidocaine mixture. No fenestration is performed.
  Interventions: Procedure: Baker's Cyst Aspiration; Drug: Steroid-Lidocaine Injection
- Arm Title: Aspiration + Steroid-Lidocaine + Fenestration (Experimental): Ultrasound-guided aspiration followed by corticosteroid-lidocaine injection and fenestration using multiple needle perforations under real-time ultrasound guidance.
  Interventions: Procedure: Baker's Cyst Aspiration; Drug: Steroid-Lidocaine Injection; Procedure: Ultrasound-Guided Fenestration

INTERVENTIONS:
Procedure: Baker's Cyst Aspiration — With the patient in the prone position, the ultrasound probe is placed transversely over the gastrocnemius-semimembranosus bursa. Under real-time ultrasound guidance, the needle is advanced while visualizing neurovascular structures to avoid injury. Aspiration of the cyst content is performed in all participants.
Drug: Steroid-Lidocaine Injection — Following aspiration, an injection mixture consisting of 1 mL betamethasone,
  1 mL of 2% lidocaine, and 1 mL of 0.9% isotonic sodium chloride is administered into the decompressed cyst cavity under ultrasound guidance.
Procedure: Ultrasound-Guided Fenestration — After aspiration, fenestration of the cyst wall is performed under ultrasound guidance. The cyst wall is punctured at a minimum of six different points using a needle to create communication with surrounding tissues and reduce recurrence. Following fenestration, the same steroid and local anesthetic mixture is administered.
  Arms: Arm Title: Aspiration + Steroid-Lidocaine + Fenestration

SUMMARY:
This study aims to evaluate whether adding a fenestration procedure to standard ultrasound-guided aspiration and corticosteroid-lidocaine injection provides additional clinical benefits for patients with symptomatic Baker's cyst associated with knee osteoarthritis. Baker's cyst is a fluid-filled swelling located behind the knee that may cause pain, stiffness, swelling, and limited mobility. Although aspiration with medication injection is commonly used to relieve symptoms, recurrence of the cyst is frequent.

Fenestration is a minimally invasive technique in which small controlled openings are created in the cyst wall under ultrasound guidance to improve internal drainage and potentially reduce recurrence. In this prospective, randomized, double-blind, controlled study, participants will be assigned to one of two groups:

1. aspiration with corticosteroid and lidocaine injection, or
2. aspiration with corticosteroid and lidocaine injection plus fenestration.

Pain, functional scores, cyst measurements, and recurrence will be assessed at follow-up visits at 2 weeks, 1 month, and 3 months. The purpose of this study is to determine whether the addition of fenestration results in better symptom improvement and lower rates of recurrence compared with standard aspiration alone.

DETAILED DESCRIPTION:
Baker's cyst, also known as a popliteal cyst, is frequently observed in patients with knee osteoarthritis and is typically associated with intra-articular pathology that increases synovial fluid production. Ultrasound-guided aspiration combined with corticosteroid-lidocaine injection is a widely used minimally invasive treatment; however, recurrence remains a significant limitation of this method.

Fenestration involves creating multiple small perforations in the cyst wall using a needle under real-time ultrasound guidance. This technique is expected to enhance communication between the cyst and surrounding tissues, promote better fluid redistribution, and reduce the likelihood of reaccumulation.

This prospective, randomized, double-blind, controlled clinical trial will enroll adult patients meeting the 2010 ACR criteria for knee osteoarthritis and demonstrating a symptomatic Baker's cyst on ultrasound. Participants will be randomized in a 1:1 ratio into two groups:

Group 1: aspiration + corticosteroid-lidocaine injection

Group 2: aspiration + corticosteroid-lidocaine injection + fenestration

All procedures will be performed by a trained physiatrist using sterile technique and real-time ultrasonography. Outcome measures include VAS pain scores, KOOS, WOMAC, Rauschning-Lindgren classification, ultrasonographic cyst dimensions, and aspirated fluid volume. Assessments will be conducted at baseline and at 2-week, 1-month, and 3-month follow-up visits.

The primary objective is to investigate whether fenestration, when added to aspiration, enhances clinical outcomes and reduces recurrence rates. Secondary objectives include evaluating functional improvements, changes in cyst size, and patient-reported symptoms. The study duration for each participant is 3 months, and the overall study is planned to be completed within 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 75 years
* Diagnosis of knee osteoarthritis according to the 2010 American College of Rheumatology (ACR) criteria
* Presence of a symptomatic Baker's cyst confirmed by ultrasonography
* Ability to understand study procedures and provide written informed consent
* Sufficient intellectual and social capacity to comply with study visits and follow-up requirements

Exclusion Criteria:

* Presence of inflammatory arthritis, septic arthritis, crystal arthropathy, or secondary causes of knee osteoarthritis
* Kellgren-Lawrence grade 4 knee osteoarthritis
* Active systemic infection
* History of malignancy
* Intra-articular knee injection within the past 3 months
* Knee trauma within the past 3 months
* History of knee surgery
* Contraindications to aspiration or corticosteroid injection (e.g., local infection, bleeding disorders, uncontrolled diabetes mellitus)
* Requirement to continue medications for inflammatory arthritis
* Diagnosed psychiatric disorder that may impair study participation
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within the past 1 week
* Physical therapy applied to the knee region within the past 1 month

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Baker's Cyst Volume | Baseline, 2 weeks, 1 month, and 3 months after the intervention
  Baker's cyst volume measured by ultrasonography using three-dimensional linear measurements (height × width × depth) and calculated in cubic millimeters (mm³). Volume measurements will be compared between the two study groups (Aspiration + Steroid-Lidocaine vs. Aspiration + Steroid-Lidocaine + Fenestration). All measurements will be performed by a blinded physician using a 7-13 MHz linear transducer. Lower values indicate a reduction in cyst size.

SECONDARY OUTCOMES:
Change in Pain Severity (NRS Score) | Baseline, 1 hour post-procedure, 2 weeks, 1 month, 3 months.
  Pain severity will be assessed using the Numeric Rating Scale (NRS; 0-10), where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Pain levels will be recorded at each follow-up visit, and changes over time will be compared between the two study groups.
Change in Rauschning-Lindgren Classification (RLC) | Baseline, 2 weeks, 1 month, 3 months.
  Clinical severity of Baker's cyst-related knee symptoms assessed using the Rauschning-Lindgren Classification, a 4-grade clinical scale ranging from Grade 0 to Grade 3. Grade 0 indicates no swelling, pain, limitation of range of motion, instability, or functional restriction. Grade 1 represents mild symptoms such as slight swelling or discomfort after strenuous activity with minimal functional limitation.
  Grade 2 corresponds to moderate swelling and pain following moderate exertion, with measurable limitation of knee range of motion and reduced participation in physical activities. Grade 3 reflects severe symptoms, including marked swelling, pain at rest or interfering with activities of daily living, significant limitation of knee motion, instability, and inability to participate in work or sports activities.
  Higher grades indicate greater clinical severity of symptoms.
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 2 weeks, 1 month, 3 months.
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) consists of five subscales: Pain (9 items), Symptoms (7 items), Activities of Daily Living (17 items), Sport and Recreation Function (5 items), and Knee-related Quality of Life (4 items).Each item is scored on a 5-point Likert scale from 0 to 4. Raw subscale scores are calculated by summing the item scores within each subscale and are subsequently transformed to a 0-100 scale using the standard KOOS transformation formula, where 0 represents extreme knee problems and 100 represents no knee problems.
  The KOOS total score is calculated as the arithmetic mean of the five normalized subscale scores. Higher total scores indicate better knee-related symptoms, function, and quality of life.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 2 weeks, 1 month, 3 months.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a disease-specific, patient-reported outcome measure consisting of 24 items grouped into three subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items).
  Each item is scored on a 5-point Likert scale ranging from 0 (none) to 4 (extreme). Raw subscale scores are calculated by summing the item scores within each subscale, with maximum possible scores of 20 for Pain, 8 for Stiffness, and 68 for Physical Function, resulting in a total raw score ranging from 0 to 96.
  For analysis, raw scores are summed to generate the WOMAC total score. Higher total scores indicate worse pain, stiffness, and physical dysfunction related to knee osteoarthritis.
Baseline OMERACT Ultrasound Score | Baseline
  Baseline knee ultrasound assessment will be performed according to the OMERACT (Outcome Measures in Rheumatology) ultrasound definitions for knee osteoarthritis.
  Synovitis will be assessed in the suprapatellar and medial/lateral parapatellar recesses using standardized longitudinal and transverse scanning planes and graded from Grade 0 to Grade 3, where higher grades indicate greater synovial distension by abnormal hypoechoic or anechoic material.
  Synovial hypertrophy will be graded from Grade 0 to Grade 1 based on the presence of non-displaceable intra-articular tissue. Joint effusion will be evaluated in the parapatellar recesses and graded as Grade 0 (absent) or Grade 1 (present). Power Doppler signal will be recorded as present or absent.
  Baseline structural findings including cartilage damage (Grade 0-3), meniscal extrusion (Grade 0-2), and osteophytes (Grade 0-3) will be documented. Higher grades indicate more severe pathology.
Change in Kellgren-Lawrence (K-L) Grade | Baseline only
  Radiographic severity of knee osteoarthritis will be assessed using the Kellgren-Lawrence (K-L) classification based on standard anteroposterior knee radiographs. The K-L grading system ranges from Grade 0 to Grade 4, where Grade 0 indicates no radiographic features of osteoarthritis; Grade 1 indicates doubtful joint space narrowing with possible osteophyte formation; Grade 2 indicates definite osteophytes with possible joint space narrowing; Grade 3 indicates multiple osteophytes, definite joint space narrowing, sclerosis, and possible bony deformity; and Grade 4 indicates large osteophytes, marked joint space narrowing, severe sclerosis, and definite bony deformity.
  Higher grades indicate more severe radiographic osteoarthritis. Baseline K-L grade will be used for descriptive and subgroup analyses, as structural radiographic change is not expected during short-term follow-up.
Change in Cyst Characteristics on Ultrasound | Baseline, 2 weeks, 1 month, 3 months.
  Baker's cyst morphology will be classified as simple or complex based on ultrasound appearance. A simple cyst is defined as an anechoic, unilocular structure without internal septations or echogenic material, whereas a complex cyst is defined by the presence of internal septations, echogenic contents, wall thickening, or irregular morphology.
  Changes in cyst complexity over time will be compared between the two study groups.
Aspirated Fluid Volume | During the procedure (single time point).
  Total volume of aspirated Baker's cyst fluid measured in milliliters (mL) during the procedure. Higher volumes indicate greater cyst content.
Change in Ultrasound Effusion Grade (OMERACT) | Baseline, 2 weeks, 1 month, and 3 months
  Joint effusion assessed by ultrasonography using the OMERACT semiquantitative grading system for knee osteoarthritis, ranging from Grade 0 to Grade 1. Grade 0 indicates no effusion, while Grade 1 indicates the presence of abnormal hypoechoic or anechoic intra-articular fluid that is displaceable and compressible and does not exhibit Power Doppler signal.
  Changes in effusion grade over time will be compared between the two study groups. Higher grades indicate greater joint effusion.

OTHER OUTCOMES:
Post-Procedure Pain Change (Short-Term Response) | Baseline and 1 hour after the procedure.
  Immediate post-procedural pain assessed using the Numeric Rating Scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores indicate worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: TUTKU NAZ BULUT, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant-level data will not be shared. Study results will be reported in aggregated form in a manner that does not allow identification of individual participants.

REFERENCES:
- [Background] Kim JM, Kang S, Yoon JS. Association of complicated Baker's cysts with knee pathologies as compared to simple Baker's cysts. Medicine (Baltimore). 2024 Jun 7;103(23):e38407. doi: 10.1097/MD.0000000000038407. PMID 38847688
- [Background] Mortada M, Amer YA, Zaghlol RS. Efficacy and Safety of Musculoskeletal Ultrasound Guided Aspiration and Intra-Lesional Corticosteroids Injection of Ruptured Baker's Cyst: A Retrospective Observational Study. Clin Med Insights Arthritis Musculoskelet Disord. 2020 Nov 10;13:1179544120967383. doi: 10.1177/1179544120967383. eCollection 2020. PMID 33223862
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Ferdousi A, Islam MA, Begum M, Debnath MR, Shapla SP, Saha T, Biswas R, Ferdouse F, Rahman MA. Diagnostic Value of Ultrasonography in Determination of Knee Joint Pathologies with Comparison to MRI. Mymensingh Med J. 2024 Oct;33(4):989-995. PMID 39351715
- [Background] Bandinelli F, Fedi R, Generini S, Porta F, Candelieri A, Mannoni A, Innocenti M, Matucci Cerinic M. Longitudinal ultrasound and clinical follow-up of Baker's cysts injection with steroids in knee osteoarthritis. Clin Rheumatol. 2012 Apr;31(4):727-31. doi: 10.1007/s10067-011-1909-9. Epub 2011 Dec 27. PMID 22200813
- [Background] Chen CK, Lew HL, Liao RI. Ultrasound-guided diagnosis and aspiration of Baker's cyst. Am J Phys Med Rehabil. 2012 Nov;91(11):1002-4. doi: 10.1097/PHM.0b013e318269d95b. No abstract available. PMID 22955026
- [Background] Oo WM, Linklater JM, Bennell KL, Pryke D, Yu S, Fu K, Wang X, Duong V, Hunter DJ. Are OMERACT Knee Osteoarthritis Ultrasound Scores Associated With Pain Severity, Other Symptoms, and Radiographic and Magnetic Resonance Imaging Findings? J Rheumatol. 2021 Feb;48(2):270-278. doi: 10.3899/jrheum.191291. Epub 2020 May 15. PMID 32414954
- [Background] Acebes JC, Sanchez-Pernaute O, Diaz-Oca A, Herrero-Beaumont G. Ultrasonographic assessment of Baker's cysts after intra-articular corticosteroid injection in knee osteoarthritis. J Clin Ultrasound. 2006 Mar-Apr;34(3):113-7. doi: 10.1002/jcu.20210. PMID 16547992
- [Background] Smith MK, Lesniak B, Baraga MG, Kaplan L, Jose J. Treatment of Popliteal (Baker) Cysts With Ultrasound-Guided Aspiration, Fenestration, and Injection: Long-term Follow-up. Sports Health. 2015 Sep-Oct;7(5):409-14. doi: 10.1177/1941738115585520. Epub 2015 May 5. PMID 26502415
- [Background] Abate M, Di Carlo L, Di Iorio A, Salini V. Baker's Cyst with Knee Osteoarthritis: Clinical and Therapeutic Implications. Med Princ Pract. 2021;30(6):585-591. doi: 10.1159/000518792. Epub 2021 Aug 2. PMID 34348320